CLINICAL TRIAL: NCT07331493
Title: Follicular Size and Oocyte Retrieval in ICSI Cycle : Establishing a Minimum Predictive Threshold. A Prospective Cohort Study
Brief Title: Establishing a Minimum Predictive Threshold Follicular Size and Oocyte Retrieval in ICSI Cycle
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Rashad Mahmoud Mostafa, Dr, Assiut University
Other Study IDs: Follicular size and ICSI
Record Dates: First submitted 2025-11-21; First posted 2026-01-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Female Infertility
Keywords: ICSI; Follicular size; Oocyte Retrieval; Oocyte yield; assisted reproduction
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICSI observational Cohort: Participants will undergo standard ICSI procedures. Follicle size and number will be measured during ovarian stimulation; and oocyte yield will be see corded at retrieval. No additional interventions will be performed. The study aims to evaluate the predictive relationship between follicle characteristics and Oocyte yield

SUMMARY:
This study uses number and size of ovarian follicles on the day of ovulation trigger as key determinants for oocytes yield to optimize outcomes in IVF and ICSI Protocols

DETAILED DESCRIPTION:
Accurate prediction of oocyte yield is a key factor in optimizing outcomes of in vitro fertilization (IVF) and intracytoplasmic sperm injection (ICSI) cycles. Follicle number and follicle diameter measured on the day of ovulation trigger are known to be strongly associated with oocyte retrieval and oocyte maturity. Larger follicles are more likely to yield mature (metaphase-II) oocytes, while smaller follicles contribute less consistently to oocyte yield.

Despite the established association between follicular size and oocyte maturity, there is currently no standardized clinical model that estimates the minimum expected number of retrieved oocytes based on the distribution of follicle diameters on the trigger day. Most existing studies focus on average outcomes rather than providing a practical tool to estimate the lowest anticipated oocyte yield for individual patients.

This study aims to estimate the minimum number of oocytes retrieved based on the number and diameter of ovarian follicles measured on the day of ovulation trigger. By developing a predictive approach based on follicular size distribution, this study seeks to support clinical decision-making, optimize trigger timing, and improve patient counseling regarding realistic expectations of oocyte yield.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 to 35 years undergoing ICSI.
* at least four follicles above 15 mm in diameter on the day of trigger
* Downregulation using either GNRH antagonist or agonist protocol
* Provision of written ,informed consent
* BMI 18 to 35 kg per meter square

Exclusion Criteria:

* anticipated poor responder, according to Bologna criteria
* cycle canceled prior to retrieval or without trigger administration
* Oocyte cryoperservation cycles or natural IVF cycles
* presence of ovarian pathology affecting the follicular assessment (endometriosis,cysts )

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female participants are eligible because the study focuses on Oocyte retrieval during ICSI, which is a procedure performed in women
Study Population: Female participants aged 18 to 35 years undergoing ICSI
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Total number of oocytes retrieved per participant during an ICSI cycle | From the start of controlled ovarian stimulation until the day of oocyte retrieval, assessed at oocyte retrieval (approximately 10-14 days after stimulation initiation and 34-36 hours after ovulation trigger).
  The total number of oocytes retrieved will be recorded for each participant. Follicular number and mean follicular diameter will be measured by transvaginal ultrasound during ovarian stimulation, and their association with oocyte yield will be analyzed to determine minimum predictive thresholds for successful oocyte retrieval.

SECONDARY OUTCOMES:
Oocyte yield stratified by follicle size category and age group | From the start of controlled ovarian stimulation until the day of oocyte retrieval, assessed at oocyte retrieval (approximately 10-14 days after stimulation initiation and 34-36 hours after ovulation trigger).
  The total number of oocytes retrieved per participant will be recorded and analyzed according to follicle size categories on the day of ovulation trigger. Participants will be stratified into predefined age groups (18-29 years and 30-35 years), and oocyte yield per follicle size category will be compared between age groups.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Ahmed Makhlouf, MD, Study Chair — Assiut University; Ahmed Abo-Elfadle, MD, Study Chair — Assiut University; Ahmed Mohamed Abo Elhasan Morsy, MD, Study Chair — Assiut University
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
No plan to share individual participant data is currently in place for this study

REFERENCES:
- See also: This website provides the official ESHRE guidelines on a Varian stimulation, follicle monitoring and IVF and ICSI protocols, including definitions of poor ovarian response, which informed the design of this study — http://www.eshre.eu/guidelines